CLINICAL TRIAL: NCT04782752
Title: Non-ablative Oligofractionated Radiation Therapy Before Surgical Transplantation As Radiovaccination
Acronym: NORTh STAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marc de Perrot (Other)
Responsible Party: Sponsor-Investigator, Marc de Perrot, Thoracic Surgeon, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-5902
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Transplant-Related Lung Cancer

STUDY DESIGN:
Intervention Model Description: 3+3 radiation dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Radiation (Experimental): Patients will be differentiated into 4 groups:
  1. Patients with end-stage interstitial lung disease (ILD) and suspected stage I (up to 4 cm) primary lung cancer
  2. Patients with end-stage lung disease other than ILD (e.g. emphysema/COPD, cystic fibrosis and pulmonary hypertension) and suspected stage I (up to 4 cm) primary lung cancer
  3. Patients with multifocal primary lung cancer (e.g. multifocal adenocarcinoma) in the absence of nodal metastasis and distant metastasis.
  4. Patients with isolated pulmonary metastasis in the absence of other sites of malignancy (primary and metastatic).
  For this study, different doses will be used for each different group depending on their tumour size. The first 3 patients will start with a dose of 4 Gy, for the ILD group, or 8 Gy, for the non ILD group. The doses are then increased incrementally until the dose limiting toxicity is reached.
  Interventions: Radiation: Radiation: Varying Doses of RT

INTERVENTIONS:
Radiation: Radiation: Varying Doses of RT — 3+3 radiation dose escalation model to see the maximum tolerated dose

SUMMARY:
This is a prospective phase I study to determine the safety and feasibility of non-ablative oligofractionated radiation therapy (NORT) before lung transplantation for patients with underlying pulmonary malignancy. We hypothesize that heterogeneous dose distributions could generate a vaccination effect against the tumor by creating anti-tumoral immune response in the body and these patients may be immunized against their tumor which could reduce the risk of cancer recurrence after transplantation despite the anti-rejection medications required for the transplantation.

DETAILED DESCRIPTION:
This study is designed to deliver short courses of radiation to the pulmonary malignancy followed by resection of the radiated tumor at the time of transplant.

The study is a 3+3 phase 1 study with incremental dose of radiation to determine the maximum tolerated dose (MTD). Dose limiting toxicity (DLT) will be defined as grade 3+ radiation related toxicity. If one DLT is seen, then an additional 3 patients will be treated at the same dose level. If 2 or more DLT are seen at any given dose level, then the previous dose level will be defined as the MTD. A minimum of 3 patients and maximum of 18 patients will be included for the phase 1a. Due to the expected higher radiation risks in patients with end-stage ILD (group 1), these patients will be stratified separately from non-ILD patients (group 2, 3 and 4) during phase 1a. Dose tested are: 3 x 400 cGy, 3 x 600 cGy and 3 x 800 cGy for the ILD cohort and 3 x 800 cGy, 3 x 1000 cGy and 3 x 1200 cGy for the non-ILD cohort.

Once the MTD is determined, patients will proceed to phase 1b using the MTD determined in the phase 1a. ILD and non-ILD patients may have different MTD so two separate phase Ib cohorts will be conducted. A total of 12 patients will be included for each cohort in the phase 1b. The dose distribution will be administered using a standard homogenous dose distribution for tumors ≤2 cm, and an heterogeneous dose distribution for tumors >2 cm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients with end-stage lung disease and suspected stage I primary lung cancer based on CT and PET scan not accessible to curative treatment, including surgery and ablative SBRT.
* Patients with multifocal pulmonary malignancy, including multifocal lung adenocarcinoma, not accessible to curative treatment, including surgery and ablative SBRT.
* Patients with isolated metastases in one or both lungs after complete resection of the primary tumor in the absence of other sites of metastatic disease, not accessible to curative treatment, including surgery and ablative SBRT.
* Meet eligibility criteria for lung transplantation with the exception of the underlying malignancy.
* Subjects must be able to understand the potential risks and benefits of the study and must be able to read and provide written, informed consent for the study.

Exclusion Criteria:

* Age < 18
* Mediastinal nodes metastasis demonstrated on EBUS-TBNA
* Distant metastasis demonstrated on PET scan or brain imaging.
* Failure to provide informed consent
* Previous thoracic radiation resulting in significant mediastinal or chest wall overlap precluding re-irradiation
* Any other medical condition that, in the opinion of the multidisciplinary team, may interfere with the subject's participation or compliance with the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose for Radiation | Up to four years
  AEs will be graded by CTCAE. Maximum tolerated dose is the dose level do not result in fatal injury (grade 5 lung toxicity) or life-threatening or fatal treatment related toxicity (grade 4+).
  Safety will be determined by the absence of grade 3 or greater (G3+) complications related to radiation and the feasibility to list patients for transplantation one week after the end of radiation will be determined.

SECONDARY OUTCOMES:
Patient Morbidity | Up to four years
  NCI common toxicity scale
Local recurrence | Up to four years
  Documented radiographically

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No